CLINICAL TRIAL: NCT02016820
Title: Effect of Proton Pump Inhibitors on the Colonic Microbiome in Children
Brief Title: Effect of Acid Suppression Medication on Pediatric Microbiome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Julian A Abrams, MD, Professor of Medicine and Epidemiology, Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAM9955
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium Difficile Infection; Proton Pump Inhibitors; Histamine-2 Receptor Antagonists; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Clostridium Infections; Gastroesophageal Reflux | interventions — Omeprazole; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (suspension) (Experimental): Open-label, with all subjects receiving omeprazole
  Interventions: Drug: Omeprazole (suspension)
- Lifestyle Modification (Other): Treated with lifestyle modification (upright feeding, smaller meals, elevation of the head of the bed, etc.)
  Interventions: Other: Lifestyle Modification

INTERVENTIONS:
Drug: Omeprazole (suspension) — 1 mg/kg/day
  Other Names: As above
  Arms: Omeprazole (suspension)
Other: Lifestyle Modification — Standard lifestyle modification: small meals, upright feeding, elevation of the head of the bed
  Arms: Lifestyle Modification

SUMMARY:
The colonic microbiome is essential in health and disease, and is highly dynamic during the first several years of life. Proton pump inhibitors (PPIs) and histamine-2 receptor antagonists (H2RAs) are widely used in children, but the effects of PPIs and H2RAs on the pediatric colonic microbiome are unknown. This study will determine whether acid suppression with these medications affects the microbiome of otherwise healthy children who are prescribed acid suppression for gastroesophageal reflux disease (GERD), and determine the duration and magnitude of microbiome changes.

DETAILED DESCRIPTION:
Otherwise healthy children age 0-4 years old who are being considered for acid suppressive therapy for GERD will be eligible for this study. Subjects donate samples before and after being treated with PPIs or H2RAs (must donate at least 2 baseline pre-PPI samples to be eligible for final analysis). 30 total children who complete the study (anticipated 10 who receive lifestyle modification and 20 who receive PPIs or H2RAs). All children will donate 6 stools on or about weeks 0, 4, 12, 20, 38, and 64. The primary outcome will be a significant change in the overall diversity of the colonic microbiome after 8 weeks of PPIs or H2RAs (i.e., from week 12 to week 4), compared to after 4 weeks of lifestyle management.

ELIGIBILITY:
Inclusion Criteria:

* Zero to 4 years old
* Being considered for PPI or H2RA treatment for refractory GERD
* Parent is able to give informed consent

Exclusion Criteria:

* Prevalent C. difficile infection (excluded via stool PCR at week 0)
* Use of systemic antibiotics within the past 90 days
* Use of acid suppression medications within the past 90 days (antacids allowed if none within the last 7 days)
* Increased risk for fracture due to vitamin D deficiency or other causes
* Chronic gastrointestinal disease (e.g. inflammatory bowel disease, celiac disease, microscopic colitis, malabsorptive conditions, short gut syndrome)
* Congenital deficiency in immunity (e.g., such as IgA deficiency)
* Cystic fibrosis
* Significant dynamic or uncontrolled comorbidity such as HIV or malignancy
* Use of medications with potential interaction with PPIs

Ages: 0 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian S Abrams, MD, MS, Principal Investigator — Columbia University; Daniel E Freedberg, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omeprazole (Suspension) | Lifestyle Modification
Started | 3 | 4
Completed | 1 | 0
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omeprazole (Suspension) | Lifestyle Modification | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Fecal Microbiome Diversity, Assessed by Bray-Curtis Index Comparing Those Who Received Acid Suppression Medications to Those Who Received Lifestyle Modifications
Time Frame: From week 12 to week 4
Population: Zero participants analyzed as only 1 participant completed. Data was not analyzed and is not included here to protect the confidentiality of this one participant.
Arm/Group | Omeprazole (Suspension) | Lifestyle Modification
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Subjects Eating High Fiber Diet
Description: At each study visit, we will assess the effects of longterm diet on the microbiome by using the Harvard-Willett Food Frequency Questionnaire. Using this data, we will classify each subject as low vs high fiber.
Time Frame: Up to Week 64
Population: as for outcome 1
Arm/Group | Omeprazole (Suspension) | Lifestyle Modification
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 64 weeks
Arm/Group | Omeprazole (Suspension) | Lifestyle Modification
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes